CLINICAL TRIAL: NCT05829733
Title: 6-month Evaluation of the Efficacy and Safety of Synolis VA 80/160 in the Treatment of Symptomatic Hip Osteoarthritis
Brief Title: 6-month Efficacy and Safety of Synolis VA 80/160 in Hip Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aptissen SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMCF A-SYN400 Hip
Record Dates: First submitted 2023-03-20; First posted 2023-04-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Osteoarthritis; Hip osteoarthritis; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYNOLIS VA 80/160 (Experimental): Single guided intra-articular injection of SYNOLIS VA 80/160
  Interventions: Device: SYNOLIS VA 80/160

INTERVENTIONS:
Device: SYNOLIS VA 80/160 — SYNOLIS VA 80/160 (hyaluronic acid 80 mg, sorbitol 160 mg)

SUMMARY:
Multicenter, independent study of Synolis VA 80/160 over a period of 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Patient with osteoarthritis of the hip. The diagnosis is based on the following criteria:
* Treated hip pain: Oxford score ≥ 21/60,
* Kellgren-Lawrence positive X-ray stage: II - III (inclusion radiograph dated no more than 6 months before the inclusion visit),
* Symptoms related to osteoarthritis of the hip for at least 2 months,
* Failure of treatments (i.e., inadequate or ineffective response to analgesics and/or NSAIDs or intolerance to NSAIDs or low-grade opioids (leaving an OXFORD score ≥ 21/60),
* Informed consent form signed by the patient,
* The patient has never had a visco supplement injection or corticosteroid injection in the hip to be treated (or more than 6 months old).

Exclusion Criteria:

* Pregnancy,
* Participation in another clinical trial,
* Skin lesion near the injection site,
* Recent or old infection of the affected joint,
* Patient with a programmed arthroplasty,
* Patient with a pathology that makes decision-making impossible,
* The patient must not have undergone non-prosthetic hip-conserving surgery such as osteotomy or arthroscopy less than 12 months old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evolution of the Oxford Hip Score (OXFORD 12) | 6 months (M6)
  Oxford Hip Score (OXFORD 12) composed of 12 questions measuring pain and hip function. Question includes 5 possible answers corresponding to a value from 1 to 5, with 5 representing the highest level of severity, and 1, the total or almost total absence of symptoms.

SECONDARY OUTCOMES:
Evolution of the Oxford Hip Score (OXFORD 12) | Month 3, Month 3 to Month 6
  Oxford Hip Score (OXFORD 12) composed of 12 questions measuring pain and hip function. Question includes 5 possible answers corresponding to a value from 1 to 5, with 5 representing the highest level of severity, and 1, the total or almost total absence of symptoms.
Self-assessment symptoms evolution | Month 3, Month 3 to Month 6
  7-point Likert scale (-3 to +3)
MCID Oxford Hip Score (OXFORD 12) | Month 3, Month 3 to Month 6
  Minimum clinically important difference on the Oxford Hip Score (OXFORD 12)
Hip prosthesis placement after the injection | Month 6
  Number of Participants with Hip prosthesis placement

OTHER OUTCOMES:
Safety and tolerability of SYNOLIS VA 80/160 | Month 6
  Serious adverse event occurrence

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de Rhumatologie, Hôpital Nord Franche-Comté, Belfort
  - Service de chirurgie orthopédique et traumatologie Centre Hospitalier de Dunkerque CHD, Dunkirk
  - Service d'Orthopédie II (Membre Inférieur, Chirurgie du Sport et Chirurgie Septique) Hôpital Salengro, CHRU de Lille, Lille